CLINICAL TRIAL: NCT02379442
Title: A Pilot Study of Early Treatment of Acute Graft Versus Host Disease With Bone Marrow- Derived Mesenchymal Stem Cells and Corticosteroids: Correlation of Disease Severity and Response With Biomarkers
Brief Title: Early Treatment of Acute Graft Versus Host Disease With Bone Marrow-Derived Mesenchymal Stem Cells and Corticosteroids
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150088; 15-H-0088
Record Dates: First submitted 2015-03-04; First posted 2015-03-05 (Estimated); Results first posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2017-12-13

CONDITIONS: Graft-Versus-Host Disease
Keywords: Graft-Versus-Host Disease; Corticosteroids; Mesenchymal Stromal Cell; Adoptive Cellular Therapy
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Target dose of 2 times 106 MSC/kg for up to 12 doses
  Interventions: Biological: MSC

INTERVENTIONS:
Biological: MSC — MSC are an adherent, fibroblast-like cell population found in the bone marrow. Allogeneic MSC for treatment can be grown from bone marrow aspirates or biopsies of normal donors.

SUMMARY:
Background:

- Sometimes after stem cells are transplanted, donor cells attack the recipient s cells and cause tissue damage. This is called acute graft-versus-host-disease (GVHD). Researchers want to see if bone marrow-derived mesenchymal stem cells (BMSC) can help treat GVHD. BMSC can travel in the body and help repair tissue. The BMSC in this study were grown from bone marrow from healthy volunteers.

Objectives:

- To test whether BMSC are safe to use soon after GVHD is diagnosed and to see how the body s immune system responds to BMSC.

Eligibility:

- People over 4 years old who had a stem cell transplant at NIH and now have acute GVHD. People who have had certain previous immunosuppressive therapy may be ineligible.

Design:

* Participants will be screened with medical history, physical exam, and blood tests. They will have a GVHD exam, including skin and stool tests. They must have a functioning central line.
* Participation will last 11 weeks: 4 8 weeks of cell infusions, then follow-up for the rest of the weeks.
* Up to 12 cell infusions:
* Participants will come to the clinic twice weekly.
* They will get medicine to prevent side effects (like Tylenol and Benadryl).
* BMSC will be given through a small plastic tube in an arm vein or through an IV catheter. It will last 20 60 minutes.
* Participants will be monitored for 1 hour.
* Follow-up visits: Up to twice a week, participants will have physical exam and blood tests. They may have a GVHD exam.
* Participants who have a tissue biopsy outside the study will be asked to send a sample to the study.

DETAILED DESCRIPTION:
This is a pilot study evaluating the addition of bone marrow-derived mesenchymal stem cell (BMSC) infusions to corticosteroids for the early treatment of acute graft versus host disease (GVHD). Acute GVHD is a major complication following allogeneic stem cell transplant. GVHD occurs when T-lymphocytes in the donor graft respond to signals from recipient cells and cause tissue damage. This process can lead to organ injury, increased risk of infection, and graft failure. Corticosteroids have been used as the primary therapy for acute GVHD for decades, and guidelines currently recommend their use as front line treatment. Recent prospective data from the Blood and Marrow Transplant Clinical Trials Network shows that GVHD will be cured in about half of patients with steroids alone. Patients who do not respond to steroids are considered steroid-resistant, and this is associated with much worse survival. It is possible to predict which patients will go on to have steroid-resistant GVHD by measuring the plasma concentration of the molecule called suppression of tumorigenicity 2 (ST2). BMSC infusions have been used to treat steroid-resistant acute GVHD successfully, but despite a track record of safety, little is known about the use of BMSC in the early treatment setting. The main objective of this study is to explore the feasibility of administering BMSC within 5 days of diagnosis of acute GVHD. Our study will for the first time use the ST2 biomarker to more accurately assign acute GVHD to steroid refractory or sensitive, and explore changes in ST2 and other biological markers of BMSC function and their correlation with clinical response. In the process of this study, we will assess the safety and feasibility of early treatment according to our regimen, obtain estimates of efficacy at important GVHD therapy time points, and determine if treatment with BMSC can prevent the progression of GVHD in patients with high risk of GVHD progression as measured by biomarkers.

The Cell Processing Section of the Department of Transfusion Medicine at the Clinical Center NIH has developed a BMSC repository at NIH. The NIH BMSC are a third party, early passage product based on the EU manufacturing approach. The NIH BMSC cellular product was administered safely to transplant recipients with steroid-resistant acute GVHD in a phase I study (protocol 12-H-0010, IND #14596) conducted from March 2012 to October 2012 at NIH. This pilot study is a continuation of the previous study and open to allogeneic stem cell transplantation recipients at NIH (age greater than or equal to 4 yrs) with de novo acute GVHD requiring systemic therapy either directly after allogeneic transplantation or following treatment with donor lymphocyte infusion. Subjects will receive BMSC infusions (target dose of 2 times 10(6) BMSC/kg for up to 12 doses) in addition to standard upfront therapy with corticosteroids. The primary endpoint will be the proportion of patients without a treatment-related severe adverse event (TRSAE) at day +56. Responses will be assessed at day +28 and +56 from the initial diagnosis. Responses will be correlated to changes in GVHD biomarkers including ST2, Reg3a, TNFR1, and IL-6. Subjects will be enrolled at first diagnosis of acute GVHD, and the first BMSC infusion will be given within 120 hours of the first dose of corticosteroids. BMSC infusions will be given twice weekly for the first 4 weeks. Subjects with a complete response at the end of week 4 will not receive further infusions. All other subjects will receive BMSC infusions weekly for four additional weeks. Safety will be monitored continuously with a stopping rule for toxicity based on the treatment-related serious adverse event rate. Research samples will be drawn at regular intervals to explore biological correlates of response and to investigate the mechanism of action of BMSC.

ELIGIBILITY:
* INCLUSION CRITERIA:
* History of any grade acute GVHD requiring systemic therapy after allogeneic stem cell transplant or DLI.

  --Subjects must have received an allogeneic stem cell transplant at NIH and be diagnosed with acute GVHD. Acute GVHD is defined using the NIH consensus definition inclusive of classic acute (less than or equal to 100 days after transplant or DLI, presence of acute GVHD features, absence of chronic GVHD features) AND persistent/recurrent/late onset acute (> 100 days after transplant or DLI, presence of acute GVHD features, absence of chronic GVHD features). Subjects with stage I and II skin only (overall Grade I) or isolated upper gastrointestinal involvement are eligible if the treating physician deems that systemic corticosteroid treatment is indicated. Biopsy confirmation of GVHD is desirable, but not required for study entry because enrollment should not be delayed awaiting biopsy or pathology results. Patients must be diagnosed with a first episode of acute GVHD requiring systemic corticosteroids and associated with preceding administration of a cellular therapy including stem cells and donor lymphocyte infusion. Patients who were treated for GVHD associated with another cellular therapy product (e.g. prior allogeneic transplant or DLI) will be allowed into the study.
* Previous immunosuppressive therapy

  * The patient must have received no systemic immune suppressive therapy for treatment of new acute GVHD (e.g. pentostatin, etanercept, denileukin difitox, etc.), except for a maximum 120 hours prior corticosteroid therapy. This does not include immune suppressive therapy for GVHD prophylaxis (e.g. calcineurin inhibitor, sirolimus, MMF, etc.). It is expected that most patients will be receiving GVHD prophylaxis as part of their transplant regimen, thus patients developing acute GVHD while on GVHD prophylaxis will still be considered eligible. Concurrent or addition of locally-acting steroid therapy (skin creams, oral budesonide, or any other locally-acting steroid preparation) is allowed.
  * There is one exception to the above stipulations: Use of the oral medication MMF (in addition to systemic corticosteroids) for the treatment of acute GVHD will be allowed. MMF is commonly given early in the treatment of acute GVHD, but it has not been shown to improve outcomes compared to steroids alone in a randomized, prospective study; therefore, treatment with MMF will not exclude patients from BMSC treatment.
* Age: Age greater than or equal to 4 years old will be allowed.
* Birth control: Subjects of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while they are being treated on this study.
* Informed consent: Signed informed consent and/or assent is required. Assent and educational materials will be provided to, and reviewed with, patients under the age of 18. The informed consent process will begin at recognition of patient eligibility.

EXCLUSION CRITERIA:

* Breast feeding or pregnant females (due to unknown risk to fetus or newborn).
* Known allergy to gentamicin.

Ages: 4 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-02-23; Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sawa Ito, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Holtan SG, Pasquini M, Weisdorf DJ. Acute graft-versus-host disease: a bench-to-bedside update. Blood. 2014 Jul 17;124(3):363-73. doi: 10.1182/blood-2014-01-514786. Epub 2014 Jun 9. PMID 24914140
- [Background] Kersting S, Koomans HA, Hene RJ, Verdonck LF. Acute renal failure after allogeneic myeloablative stem cell transplantation: retrospective analysis of incidence, risk factors and survival. Bone Marrow Transplant. 2007 Mar;39(6):359-65. doi: 10.1038/sj.bmt.1705599. PMID 17342159
- [Background] Martin PJ, Rizzo JD, Wingard JR, Ballen K, Curtin PT, Cutler C, Litzow MR, Nieto Y, Savani BN, Schriber JR, Shaughnessy PJ, Wall DA, Carpenter PA. First- and second-line systemic treatment of acute graft-versus-host disease: recommendations of the American Society of Blood and Marrow Transplantation. Biol Blood Marrow Transplant. 2012 Aug;18(8):1150-63. doi: 10.1016/j.bbmt.2012.04.005. Epub 2012 Apr 14. PMID 22510384

RESULTS

PARTICIPANT FLOW:
Groups:
- BMSC: Bone Marrow-Derived Mesenchymal Stem Cells and Corticosteroids. Target dose of 2 times 10e^6 MSC/kg for up to 12 doses
Period: Overall Study
Arm/Group | BMSC
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BMSC
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Without a Treatment Related Severe Adverse Event
Description: The number of subjects without a treatment related severe adverse event (TRSAE) within 56 days of treatment.
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | BMSC
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 56 days
Arm/Group | BMSC
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
One subject completed the protocol, and the FDA placed the study on hold due to NIH operational issues. Since the cellular product of bone-marrow derived mesenchymal stem cells is no longer available, the protocol was terminated on December 13, 2017.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT02379442/Prot_SAP_000.pdf